CLINICAL TRIAL: NCT00789841
Title: Gastrointestinal Motility in Patients With Neuroendocrine Tumors-Effects of Sandostatin LAR
Brief Title: Gastrointestinal Motility in Patients With Neuroendocrine Tumors
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Novartis (Industry); The Danish Medical Research Council (Other)
Responsible Party: Henning Grønbæk, M.D., Ph.D., Medical Department V, Aarhus University Hospital
Other Study IDs: M-20080121
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-10

CONDITIONS: Neuroendocrine Tumor
Keywords: Neuroendocrine tumor; Carcinoid syndrome; Motility; Transit time
MeSH Terms: conditions — Neuroendocrine Tumors; Serotonin Syndrome

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Blood samples wich are destroyed after analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with NET and diarrhea.
  Interventions: Device: Magnetic Tracking System (MTS) and radio-opaque markers

INTERVENTIONS:
Device: Magnetic Tracking System (MTS) and radio-opaque markers — MTS: A small magnetic pill (6x15mm) is swallowed by the patient and the movement of this pill is registered by a sensor (coordinates x,y,z angles θ, φ) and depicted af graphs on a computer screen. For determination of GITT a capsule containing 10 radio-opaque markers is ingested every day for six days, on day seven an abdominal x-ray is performed.

SUMMARY:
We will study the total gastrointestinal transit time (GITT), gastric emptying and small intestine motility in NET patients before and after treated with somatostatin analogues and compare these to healthy subjects. For this we will use radio-opaque markers and the newly developed Motility Tracking System (MTS).

Hypothesis: Patients with NET and carcinoid syndrome have decreased GITT, gastric emptying and small bowel transit time and an increase in phase III MMC activity compared to healthy subjects. Treatment with somatostatin analogues increase transit times and decrease phase III MMC activity and improves the clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

* NET confirmed by histology
* Diarrhea, (at least 3 loose or watery bowel movements per day) as part of carcinoid syndrome.
* Newly referred patients without previous somatostatin analogue treatment or
* NET patients who are pausing somatostatin analogue treatment due to other treatment or examination.

Exclusion Criteria:

* Subjects unable to understand the information
* Severe diabetes with late complications or known metabolic disorder
* Inflammatory bowel disease
* Known clinically significant stenosis of the bowel
* Bile acid malabsorption due to intestinal surgery
* Small bowl bacterial overgrowth

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We are scheduling 12 subjects (30-80 years of age) with NET and carcinoid syndrome with diarrhea. Patients are recruited through the Department of Medicine V, Aarhus University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2008-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal transit time in NET patients | End of the study

SECONDARY OUTCOMES:
Gastric emptying in NET patients | End of the study
Small intestinal transit time | End of the study
Small intestinal velocity | End of the study
Changes in carcinoid symptoms and biomarkers | End of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Analfysiologisk afsnit, Aarhus University Hospital, Tage Hansensgade, entrance 11A, Aarhus, Aarhus, Denmark